CLINICAL TRIAL: NCT00628589
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Multi-Dose Efficacy and Safety Study of Staccato® Loxapine for Inhalation in Schizophrenic Patients With Agitation
Brief Title: Staccato Loxapine in Agitated Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-004-301
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2008-06

CONDITIONS: Patients With Schizophrenia and Acute Agitation
Keywords: schizophrenia, agitation, inhaled loxapine, ADASUVE
MeSH Terms: conditions — Schizophrenia; Psychomotor Agitation | interventions — Loxapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Inhaled Loxapine 5 mg (Experimental): Inhaled Loxapine 5 mg, may repeat x 1 or 2 after 2 hours
  Interventions: Drug: Inhaled loxapine 5 mg
- Inhaled Loxapine 10 mg (Experimental): Inhaled Loxapine 10 mg, may repeat x 1 or 2 after 2 hours
  Interventions: Drug: Inhaled loxapine 10 mg
- Inhaled placebo (Placebo Comparator): Inhaled Loxapine placebo, may repeat x 1 or 2 after 2 hours
  Interventions: Drug: Inhaled placebo

INTERVENTIONS:
Drug: Inhaled loxapine 5 mg — Inhaled loxapine 5 mg
  Other Names: ADASUVE
  Arms: Inhaled Loxapine 5 mg
Drug: Inhaled loxapine 10 mg — Inhaled loxapine 10 mg
  Other Names: ADASUVE
  Arms: Inhaled Loxapine 10 mg
Drug: Inhaled placebo — Inhaled placebo
  Arms: Inhaled placebo

SUMMARY:
Phase 3 safety and efficacy study of Staccato Loxapine in the treatment of acute agitation in schizophrenic patients

DETAILED DESCRIPTION:
This is an in-clinic, multi-center, randomized, double-blind, placebo-controlled study of 2 dose levels of Staccato Loxapine, 5 and 10 mg. Patients may receive up to 3 doses of study drug in a 24-hour period, depending on their clinical status. The primary endpoint is the change from baseline in the PANSS (Positive and Negative Symptom Scale) Excited Component (also known as PEC) score, performed at 2 hours after the first dose.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients with schizophrenia and acute agitation

Exclusion Criteria:

* Agitation caused primarily by acute intoxication
* History of drug or alcohol dependence
* Treatment with benzodiazepines or other hypnotics within 4 hours prior to study drug administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Fishman, MD, Study Director — Alexza Pharmaceuticals, Inc.
Locations (1):
- Atlanta Center for Medical Research, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

REFERENCES:
- [Background] Lesem MD, Tran-Johnson TK, Riesenberg RA, Feifel D, Allen MH, Fishman R, Spyker DA, Kehne JH, Cassella JV. Rapid acute treatment of agitation in individuals with schizophrenia: multicentre, randomised, placebo-controlled study of inhaled loxapine. Br J Psychiatry. 2011 Jan;198(1):51-8. doi: 10.1192/bjp.bp.110.081513. PMID 21200077
- [Derived] Zeller S, Zun L, Cassella JV, Spyker DA, Yeung PP. Response to inhaled loxapine in patients with schizophrenia or bipolar I disorder: PANSS-EC responder analyses. BJPsych Open. 2017 Nov 10;3(6):285-290. doi: 10.1192/bjpo.bp.117.005363. eCollection 2017 Nov. PMID 29163985

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 24 centers - all in the US. Patients recruited for screening were admitted to a hospital or research unit with acute agitation, and were being treated for chronic underlying schizophrenia.
Pre-assignment Details: During the Pre-treatment Period, agitated schizophrenic patients were screened for inclusion in the study. This period lasted until the evaluations were begun.
Period: Overall Study
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg
Started | 115 | 116 | 113
Completed | 114 | 114 | 110
Not Completed | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg | Total
Number analyzed (Participants) | 115 | 116 | 113 | 344
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 115 | 116 | 113 | 344
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (9.45) | 43.2 (10.24) | 42.2 (9.82) | 43.1 (9.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 29 | 27 | 91
  Male | 80 | 87 | 86 | 253
Region of Enrollment [Number; unit: participants]
  United States | 115 | 116 | 113 | 344

OUTCOME MEASURES:

1. Primary Outcome: Change in PANSS-EC From Baseline
Description: The Positive and Negative Syndrome Scale-Excited Component (PANSS-EC) comprises 5 items associated with agitation: poor impulse control, tension, hostility, uncooperativeness, and excitement; each scored 1 (min) to 7 (max). The PANSS-EC, the sum of these 5 subscales, thus ranges from 5 to 35. Individuals were eligible if they had a PANSS-EC of ≥14 (out of 35) and a score ≥4 (out of 7) on at least 1 of the 5 items.
Time Frame: Baseline and 2 hours
Population: ITT Population with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg
Number analyzed (Participants) | 115 | 116 | 112
units on a scale | -5.5 (4.92) | -8.1 (5.17) | -8.6 (4.37)
Statistical Analysis 1: Comparison: Inhaled Placebo vs Inhaled Loxapine 5 mg; Test type: Superiority — LS mean was used in the primary efficacy analysis; p = 0.0004, ANCOVA; p-values (adjusted) using Dunnett's t-test in main effects ANCOVA model
Statistical Analysis 2: Comparison: Inhaled Placebo vs Inhaled Loxapine 10 mg; Test type: Superiority; p < 0.0001, ANCOVA; p-values (adjusted) using Dunnett's t-test in main effects ANCOVA model

2. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Score
Description: Clinical Global Impression- Improvement (CGI-I) scores ranged from 1 to 7: 0=not assessed (missing), 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse.
Time Frame: Baseline and 2 hours
Population: ITT Population with LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg
Number analyzed (Participants) | 115 | 116 | 112
units on a scale | 2.8 (1.11) | 2.3 (1.24) | 2.1 (1.00)
Statistical Analysis 1: Comparison: Inhaled Placebo vs Inhaled Loxapine 5 mg; Test type: Superiority; p = 0.0015, Fisher Exact
Statistical Analysis 2: Comparison: Inhaled Placebo vs Inhaled Loxapine 10 mg; Test type: Superiority; p < 0.0001, Fisher Exact

3. Secondary Outcome: CGI-I Responders
Description: Frequency of response based on the CGI-I (defined as achieving a CGI-I score of 1 or 2 at 2 hours after administration of the inhalation)
Time Frame: Baseline and 2 hours
Population: ITT Population with LOCF
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg
Number analyzed (Participants) | 115 | 116 | 112
Participants | 41 | 66 | 75
Statistical Analysis 1: Comparison: Inhaled Placebo vs Inhaled Loxapine 5 mg; Test type: Superiority; p = 0.0015, Fisher Exact
Statistical Analysis 2: Comparison: Inhaled Placebo vs Inhaled Loxapine 10 mg; Test type: Superiority; p < 0.0001, Fisher Exact

ADVERSE EVENTS:
Time Frame: From informed consent through 30 days after last treatment
Description: AEs were recorded when identified by the study center staff or volunteered by a patient.
Arm/Group | Inhaled Placebo | Inhaled Loxapine 5 mg | Inhaled Loxapine 10 mg
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/116 | 0/113
Serious Adverse Events (participants affected / at risk) | 1/115 | 0/116 | 1/113
Other Adverse Events (participants affected / at risk) | 44/115 | 35/116 | 41/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Placebo (N=115) | Inhaled Loxapine 5 mg (N=116) | Inhaled Loxapine 10 mg (N=113)
Exacerbation of schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — A 45 year-old white male assigned to the Placebo group experienced a severe exacerbation of schizophrenia and was hospitalized.
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — A 37 year-old female assigned to the Staccato Loxapine 10-mg group had severe gastroenteritis that resulted in hospitalization. This event was reported as an SAE, was judged unrelated to study treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Placebo (N=115) | Inhaled Loxapine 5 mg (N=116) | Inhaled Loxapine 10 mg (N=113)
Dysgeusia (Gastrointestinal disorders) | 3 (3) | 10 (10) | 12 (12)
Nausea (Gastrointestinal disorders) | 6 (6) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 11 (11) | 6 (6) | 12 (12)
Headache (Nervous system disorders) | 16 (16) | 3 (3) | 3 (3)
Sedation (Nervous system disorders) | 11 (11) | 15 (15) | 12 (12)

LIMITATIONS AND CAVEATS:
Because of the need to provide informed consent, the types of patients enrolled in the study may not have been representative of the most severely agitated patients who present for emergency care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.